CLINICAL TRIAL: NCT05274139
Title: The Prospective Study of FTD Program and HD-MTX-Ara-C Program Contrast in the Treatment of PCNSL Lymphoma.
Brief Title: Treatment of Primary CNS Lymphoma ( FTD )
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mingzhi Zhang (Other)
Collaborators: Zhengzhou University (Other)
Responsible Party: Sponsor-Investigator, Mingzhi Zhang, the director of oncology department of the first affiliated hospital, Zhengzhou University
Organization: Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hnslblzlzx2017-3
Record Dates: First submitted 2017-03-10; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Primary CNS Lymphoma (PCNSL)
Keywords: primary CNS lymphoma; chemotherapy; RR; PFS; OS
MeSH Terms: interventions — Cytarabine; fotemustine; Temozolomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FTD regimen (Experimental): FTD regimen(fotemustine, temozolomide and dexamethasone),fotemustine 100mg/m2 d1 ivgtt, temozolomide 150mg/m2 d1-5 po,dexamethasone 40mg d1-5 ivgtt.Continued use to the end of chemotherapy .Every 28 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles.
  Interventions: Drug: FTD regimen
- HD-MTX-Ara-C regimen (Experimental): high-does metrotrexate 3.5g/m2 d1 ivgtt 6h,cytarabine 1g/m2 bid d2-3.Continued use to the end of chemotherapy .Every 21 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles.
  Interventions: Drug: HD-MTX-Ara-C regimen

INTERVENTIONS:
Drug: HD-MTX-Ara-C regimen — HD-MTX-Ara-C regimen high-does metrotrexate 3.5g/m2 d1 ivgtt 6h,cytarabine
  1g/m2 bid d2-3.Continued use to the end of chemotherapy .Every 21 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles
  Other Names: high-does metrotrexate and cytarabine
  Arms: HD-MTX-Ara-C regimen
Drug: FTD regimen — FTD regimen(fotemustine, temozolomide and dexamethasone),fotemustine 100mg/m2 d1 ivgtt,temozolomide 150mg/m2 d1-5 po,dexamethasone 40mg d1-5 ivgtt.Continued use to the end of chemotherapy .Every 28 days for one cycle and four cycles are required. Efficacy was evaluated every two cycles
  Other Names: fotemustine, temozolomide and dexamethasone
  Arms: FTD regimen

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of FTD regiment (fotemustine, temozolomide and dexamethasone ) for patients with primary CNS lymphoma.

DETAILED DESCRIPTION:
Primary CNS lymphoma (PCNSL) is a rare B-cell variant of non-Hodgkin lymphoma that is confined to the brain, leptomeninges, spinal cord, and eyes. The optimum treatment for patients with PCNSL remains challenging and at present there is no universally accepted therapeutic approach for patients with newly diagnosed disease. The purpose of this study is to evaluate the efficacy and safety of FTD regiment(fotemustine, temozolomide and dexamethasone)contrast with HD-MTX-Ara-C program for patients with primary CNS lymphoma.

ELIGIBILITY:
Inclusion Criteria:

Age range 14-69 years old;KPS performance status≥60 or ECOG performance status 0-2; Estimated survival time > 3 months; Histological confirmed PCNSL; None of chemotherapy contraindication;At least one measurable lesion according to RECIST;None of other serious diseases;Patients could be followed up;None of other relative treatments including the traditional Chinese medicine, immunotherapy,biotherapy except anti-bone metastasis therapy and other symptomatic treatments.

volunteers who signed informed consent.

Exclusion Criteria:

Currently undergoing chemotherapy, radiotherapy and targeted therapy (received chemotherapy within 3 weeks, received radiotherapy within 2 weeks, or has not recovered from any previous treatment of acute toxicity);Patients with uncontrolled medical problems (including active infection, uncontrolled diabetes, severe heart, liver, kidney dysfunction and interstitial pneumonia, etc.); Pregnant or lactating women;Serious medical illness likely to interfere with participation;Chemotherapy contraindication such as cachexia; patients with other malignancies previously;Serious infection;The evidence of peripheral nervous disorder or dysphrenia; patients estimated to be unsuitable by investigato

Ages: 14 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2019-03-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | up to end of follow-up-phase(approximately 24 months)
  Progression-free survival

SECONDARY OUTCOMES:
response rate | every 6 weeks,up to completion of treatment(approximately 18 weeks )
  response rate
overall survival | up to the date of death (approximately 5 years)
  overall survival
median survival time | 24 months
  median survival time

CONTACTS AND LOCATIONS:
Overall Officials: Mingzhi zhang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- Oncology Department of The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China